CLINICAL TRIAL: NCT02244216
Title: Postmarketing Surveillance Study (as Per § 67 (6) AMG [German Drug Law]) of Berotec® N 100 µg Metered-dose Inhaler in Chronic Obstructive Respiratory Tract Disease
Brief Title: Postmarketing Surveillance Study of Berotec® N 100 µg Metered-dose Inhaler in Chronic Obstructive Respiratory Tract Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 260.3178
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Metered Dose Inhalers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Obstructive Respiratory Tract Disease
  Interventions: Drug: Berotec® N 100 µg Metered-dose Inhaler

INTERVENTIONS:
Drug: Berotec® N 100 µg Metered-dose Inhaler

SUMMARY:
Study to obtain data about changing from the chlorofluorocarbon (CFC) - containing Berotec® 200 µg metered - dose inhaler to the CFC - free Berotec® N 100 µg metered - dose inhaler

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study only if they had been treated with Berotec® 200 µg metered - dose inhaler before switching to the CFC-free Berotec® N 100 µg metered - dose inhaler

Exclusion Criteria:

• Contraindications listed in the Instructions for Use/Summary of Product Characteristics for Berotec® N 100 µg metered - dose inhaler

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patinet with chronic obstructive respiratory tract disease recruited at general practitioners, pneumologists, internists
Sampling Method: Non-Probability Sample
Enrollment: 2914 (Actual)
Dates: Start 2000-04; Primary Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Change in the clinical picture of chronic obstructive airways disease on switching from Berotec® 200 µg to Berotec® N 100 µg | After 3 weeks of first drug administration

SECONDARY OUTCOMES:
Investigator assessment of efficacy on a 4-point scale | Up to 3 weeks after first drug administration
Patient assessment of efficacy on a 4-point scale | Up to 3 weeks after first drug administration
Patient assessment of tolerability on a 4-point scale | Up to 3 weeks after first drug administration
Investigator comparative overall assessment on a 4-point scale | After 3 weeks of first drug administration
Number of patients with adverse drug reactions | Up to 3 weeks after first drug administration
Number of patients who changed the concomitant medication | Up to 3 weeks after first drug administration
Number of patients who continued treatment | Up to 3 weeks after first drug administration
Number of patients who premature withdrew from the treatment | Up to 3 weeks after first drug administration